CLINICAL TRIAL: NCT04277325
Title: Efficacy of Emotionally Focused Therapy Among Spanish Speaking Couples: A Randomized Clinical Trial
Brief Title: Efficacy of Emotionally Focused Therapy Among Spanish Speaking Couples
Acronym: E(f)FECTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Brigham Young University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E(f)FECTS
Record Dates: First submitted 2020-02-11; First posted 2020-02-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Partner Relational Problems
Keywords: Emotionally Focused Therapy; Spanish Speaking couples; Couple therapy
MeSH Terms: interventions — Emotion-Focused Therapy

STUDY DESIGN:
Intervention Model Description: Couples will be randomly assigned to one of two groups: intervention or waitlist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Couples will receive 19-21 free sessions of Emotionally-Focused Therapy.
  Interventions: Behavioral: Emotionally Focused Therapy
- Waitlist (No Intervention): Couples will receive no intervention during the trial. After the trial is ended, they will be invited to participate in a weekend intervention meeting.

INTERVENTIONS:
Behavioral: Emotionally Focused Therapy — Emotionally Focused Couples Therapy (EFT) is an empirically supported, attachment-based model of couples therapy that combines experiential, systems, and attachment theories with the goal of fostering the development of safe contact, accessibility, and responsiveness in both partners.
  Arms: Intervention

SUMMARY:
70 couples (married or cohabiting) will be recruited across 5 countries (12-18 in each country: Argentina, Costa Rica, Guatemala, México, and Spain). After their entry into the study is confirmed, couples will be randomly allocated into one of two groups: intervention or control (no intervention). In each country, both groups will have equal number of couples.

Couples in the intervention group will receive 20 sessions of Emotionally Focused couple Therapy (EFT). Couples in the control group will receive no intervention during the study period (they will receive a shorter intervention after the trial is over). Participants of both groups will fill questionnaires before allocation, during the intervention period and after the intervention period.

The main outcomes will be couple attachment, couple satisfaction and dyadic adjustment.

The original timeline for the study was to start in Argentina and Guatemala in February 2020, and the remaining countries in September 2020. The study started in February 2020 for Argentina and Guatemala, but in April 2020 the process was postponed due to mobility constrains during covid-19 crisis. During these two months, the process remained in the recruitment phase. Therefore, couples were not randomly assigned. Due to an improvement in the pandemic situation, the study started in Spain in September 2021.We expect the remaining countries will start during 2022.

The study period for each couple will be around 6 months.

DETAILED DESCRIPTION:
A detailed description about the procedure of this clinical trial will be available on an open access study protocol document or paper upon request.

Some more details about therapists, supervision during treatment phase, implementation checking and research team, is offered below.

Participating therapists were chosen based on a rigorous criterion focused on excellence in the adherence to the EFT model. There therapists also had to meet the following prerequisites: (1) Meet all legal requirements necessary to practice therapy in the country and region in which the therapist is located (licensure, insurance, etc.); (2) Have a video recording device; (3) Have completed the Externship, Core Skills and at least 10 hours of EFT supervision by the 1st of June, 2019; (4) Have experience applying the EFT model in couples therapy; and (5) be a licensed therapist or actively participating in case supervision. Additionally, candidates for participating therapists must send a video of at least 20 minutes of a session of actual couples therapy recorded in the last three months, to the principal investigator (MR-G) with their application. The couple in the recording was asked for their consent to have this video be reviewed by two supervisors who are participating in the study. Each video was shared through a secure channel with Martiño Rodríguez, who then sent said video to two EFT certified therapists and/or supervisors from a list of six therapists provided by Samuel Jinich, PhD and Certified EFT Trainer. Each evaluator submitted their evaluation independently to the principle investigator. In the event that a discrepancy arose, a third evaluation was sought from a separate evaluator. In some cases, a second video was requested to resolve doubts regarding a candidate's suitability. A total of 26 therapists sent in an application to participate, of those 11 applications were considered insufficient, and 15 met the requirements of the evaluation. This application and evaluation process took place between January and September, 2019.

All sessions will be videotaped and/or audio-taped for supervision and research purposes.

Supervision of the therapy process will be offered biweekly, in an individual meeting (one therapist, one supervisor) of one hour. Participating supervisors are required to speak Spanish and to certified as a supervisor by the International Center for Excellence in Emotionally Focused Therapy; Ottawa, Canada (ICEEFT), or to be certified by ICEEFT as a therapist and actively be in the process of becoming an ICEEFT certified supervisor.

In order to ensure the therapists in this study are implementing EFT faithfully, two different procedures will be carried out. First, during the supervision meetings with participating therapists, the supervisor will review video recording segments of therapy to determine if EFT is being conducted with adherence to the model. Second, once the study ends, two independent raters will be asked to rate at least 5 sessions of each therapist's taped sessions to ensure that at least 80% of the therapists' interventions can be coded as adherent to the model.

The research team, with their relevant experience, includes the following individuals: Martiño Rodriguez-Gonzalez, Ph.D. (Principal Investigator, Certified Couple Therapist in Spain and Researcher at the Institute for Culture and Society (ICS), Universidad de Navarra, Spain), Shayne Anderson, Ph.D., (Co-Principal investigator; Associate Professor at the Brigham Young University (BYU), USA, and Psychotherapist at the BYU Comprehensive Clinic, USA), Marie-France Lafontaine, Ph.D., (Director of the Couple Research Laboratory, Full Professor at the University of Ottawa and a certified psychologist in Ontario and Quebec, Canada), Paul Greenman, Ph.D. (Full Professor and Chair of the Department of Psychoeducation and Psychology at the Université du Québec en Outaouais, and a certified psychologist in Ontario and Québec, Canada), Alfonso Osorio, Ph.D. (Associate Professor at the School of Education and Psychology and researcher at the Institute for Culture and Society, ICS, Universidad de Navarra, Spain), Jonathan Sandberg, Ph.D. (Full Professor School of Family Life at the Brigham Young University, USA), Jokin de Irala, PhD. (Associate Professor at the School of Medicine and Principal Investigator of the Research group "Educación de la afectividad y de la sexualidad humana" (EASH) at the Institute for Culture and Society, ICS, Universidad de Navarra, Spain), Patrick Steffen, Ph.D. (Full Professor in the Psychology Department at the Brigham Young University, USA), María Calatrava, Ph.D. (Researcher at the Institute for Culture and Society, ICS, Universidad de Navarra, Spain), Maria del Pilar Martínez, PhD. (Full Professor at the School of Social sciences, Department of Psychology, Universidad Pontificia Comillas, Madrid, Spain).

ELIGIBILITY:
Inclusion Criteria:

* Each couple has to be exclusive in their courtship and been living together for at least 1 year. Participants must be willing to participate in all of the study components (questionnaires, videotaping, therapy, and follow-up once therapy is finished). Each member of the relationship must speak Spanish as a native language and have lived in the country where the study is going to be conducted (Argentina, Costa Rica, Guatemala, Mexico, Spain) for at least 5 years. Couple's average score on the Dyadic Adjustment Scale (DAS; Spanier, 1976) must classify the relationship as mildly to moderately distressed (80-100).

Exclusion Criteria:

* Either partner of the couple is receiving current psychotherapeutic (psychological or psychiatric) treatment or anticipates receiving this type of treatment (not directly involved with this study) within the next 6 months.
* Either member has been previously diagnosed with any psychotic, somatoform or dissociative disorder.
* Either partner is currently taking any medication known to treat psychosis, somatoform, dissociative or psychotic disorders or is taking any psychotropic medication, has a diagnosis of a neurodevelopmental (e. g., autism spectrum disorder), neurocognitive, personality or paraphilic disorder.
* Either partner reports having been arrested or in prison in the past 3 months due to driving drunk or any other legal problem related to alcohol or other drugs, reports having been fired from her/his job due to alcohol or substance use/abuse, reports an episode (as a victim and/or perpetrator) of a sexual assault during the past 2 years, reports current physical or sexual violence in their relationship, or is currently involved in an affair which he/she will not end or requests that the affair remains secret.
* Either partner has a condition or anticipates having a condition that may make attending therapy sessions unlikely (e.g., major surgery expected in the next 3 months, or moving to a new area in the near future, etc.), is misusing/abusing drugs or alcohol, is a psychotherapist active in clinical practice and/or has a direct knowledge of the model because he/she is in training or trained in EFT.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Change in Dyadic Adjustment Scale (DAS-32 and DAS-4) | Baseline and up to 6 months
  The Dyadic Adjustment Scale (DAS; Spanier, 1976) is a 32- item measure which measures romantic relationship adjustment. Partners are asked to rate the occurrence of both relationship disagreements and positive relationship exchanges on a Likert scale from 1-5 or 1-6. Higher scores on this measure are indicative of better relationship adjustment or higher relationship satisfaction. A short version of the DAS called the DAS-4 (Sabourin, Valois, & Lussier, 2005), composed of 4 items, will also be used. The DAS-4 measure was chosen to decrease the time spent by couples completing questionnaires coinciding with their therapy sessions.
Change in Couple Satisfaction Inventory (CSI-16) | Baseline and up to 6 months
  The CSI-16 (Funk & Rogge, 2007) is a 16-item measure of relationship satisfaction. One global item uses a 7-point scale, whereas the other 15 items use a variety of response anchors, all with 6-point scales. The CSI represents the only measure of relationship satisfaction described here which was developed using item response theory. Higher scores indicate higher levels of relationship satisfaction.
Change in Experiences in Close Relationships Questionnaire (ECR-36) | Baseline and up to 6 months
  This measure contains 36 items and yields continuous scores on two attachment domains: attachment anxiety and attachment avoidance. The data collected through the ECR would contribute to this study as it would allow researchers to analyze the effect of EFT therapy on the attachment styles of clients living in Spanish speaking countries.

SECONDARY OUTCOMES:
Change in General Health Questions (Health-4) | Baseline and up to 6 months
  In this measure, respondents are asked to rate their health. Higher scores on this measure represent better health. Participants respond to these questions about general health based on a 5-point Likert scale ranging from 1 (poor) to 5 (excellent). As there are many established connections between mental health and physical health, these variables are of interest in this study so as to control for the effects of physical health or physical ailments on participant outcomes as well as an analysis of the positive effects of relationship quality increases on physical health.
Change in Patient Health Questionnaire (PHQ - 15) | Baseline and up to 6 months
  The PHQ-15 is a somatic symptom subscale which stems from the original full PHQ. The PHQ has 13 somatic and 2 psychological (fatigue, sleep problems) symptoms questions. Each item is scored from 0 (not bothered at all) to 2 (bothered a lot). Items consist of symptoms such as "stomach pain" and "headaches" (Kroenke, Spitzer & Williams, 2002).
Change in Depression Anxiety Stress Scale (DASS-21) | Baseline and up to 6 months
  The DASS 21 consists of 21 negative emotional symptoms statements/questions. Respondents rate to what extent over the past week they have experienced each symptom on a 4-point scale of severity or frequency. The DASS 21 has a depression, anxiety and stress subscale. Items on the depression subscale consist of statements like "I felt that life was meaningless." and "I felt down-hearted and blue." Items on the stress subscale consist of statements like "I felt I was rather touchy." and "I found it difficult to relax." Items on the anxiety subscale consist of statements like "I felt I was close to panic." and "I felt scared without any good reason." (Antony, Bieling, Cox, Enns, & Swinson, 1998).
Change in Sexual dissatisfaction subscale of Marital Satisfaction Inventory (SD-13) | Baseline and up to 6 months
  The Revised Marital Satisfaction inventory has 150 items which measure the type and severity of relationship distress in multiple areas of marital interaction including aggression, finances, role orientation, leisure time spent together etc. Respondents choose between a true and false response to each item. The Sexual dissatisfaction (SD-13) subscale assesses the level of dissatisfaction through statements regarding the frequency and quality of the couple's sexual activity. Items consist of statements such as "My spouse sometimes shows too little enthusiasm for sex." and "My spouse has too little regard sometimes for my sexual satisfaction." (Snyder, 1979).
Change in UCLA Loneliness Scale Revised - Short version (UCLA LS-R-8) | Baseline and up to 6 months
  The revised UCLA loneliness scale (UCLA LS-R) is a 8-item questionnaire designed to measure and detect variations in loneliness. Each item is ranked on a 4-point Likert scale ranging from "Never" to "Often". Items consists of statements like "I feel isolated from others" and "I lack companionship" (Hays & DiMatteo, 1987). As loneliness can be an indicator of relationship satisfaction and/or relationship quality, data collected through this questionnaire would allow researchers to assess for an additional element of relationship satisfaction and the impact EFT has on relationship satisfaction.
Change in Reflective functioning questionnaire (RFQ-8) | Baseline and up to 6 months
  The RFQ seeks to measure the capacity one has to understand one's own and other's feelings, goals and attitudes. It has an uncertainty subscale and a certainty subscale. This short version of the RFQ contains 8 items which are scored on a 7-point Likert scale ranging from "strongly disagree" to "strongly agree". Items consist of statements such as "People's thoughts are a mystery to me" and "I always know what I feel." This scale would provide data allowing researchers to control for individual's capacity for understanding their partner and how EFT might affect said capacity.
Change in Authoritative Parenting subscale (RELATE)-(AP-15) | Baseline and up to 6 months
  The Authoritative Parenting subscale comes from the Parenting Style and Dimensions Questionnaire Short form (PSDQ). The PSDQ is used to measure parenting styles. The authoritative parenting subscale from the short version of the PSDQ is composed of 15 items. (Olivari, Tagliabue, & Confalonieri, 2013; Oliveira et al., 2018). Items include phrases such as "I am responsive to our child's feelings or needs." and "I allow our child to give input into family rules." Responses are scored on a 5-point Likert scale ranging from "Never" to "Always" (Oliveira et al., 2018).
Change in Sleep quality (Sleep-8) | Baseline and up to 6 months
  The PROMIS sleep disturbance short form (Sleep-8) questionnaire has 8 items. Respondents are asked to assess their sleep quality over the past 7 days by responding to statements like "I had trouble sleeping." and "My sleep was refreshing." Responses are scored on a 5-point Likert Scale ranging from "Not at all" to "Very Much."
Change in The Brief Accessibility, Responsiveness, and Engagement Scale (BARE-12) | Baseline and up to 6 months
  The BARE is an instrument which measures an individual's perception of their own and their partners attachment behaviors. It measures attachment behaviors (and has 3 subscales) through assessing accessibility, responsiveness and engagement, all of which are related to secure attachment. The scale has 12 items, measuring 6 subscales (accessibility, responsiveness and engagement for both self and partner). Items are scored on a 5-point Likert scale ranging from "Never True" to "Always True." Items consist of statements such as "I am rarely available to my partner." and "I am confident my partner reaches out to me." (Sandberg, Busby, Johnson, & Yoshida, 2012).
Change in CORE Outcome Measure short form (CORE-OM-10) | Baseline and up to 6 months
  This is a client self-report questionnaire designed to be administered before and after therapy. The questionnaire is repeated after the last session of treatment; comparison of the pre-and post-therapy scores offers a measure of 'outcome' (i.e. whether or not the client's level of distress has changed, and by how much). The CORE-10 is a brief outcome measure comprising 10 items drawn from the CORE-OM which is a 34-item assessment and outcome measure. The CORE-OM has been widely adopted in the evaluation of counseling and the psychological therapies in the UK. The CORE-10 taps global distress and is, therefore, suitable for use as an initial quick screening tool and also as an outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Martiño Rodríguez-González, PhD, Principal Investigator — University of Navarra; Shayne Anderson, PhD, Principal Investigator — Brigham Young University
Locations (16):
- Argentina (4):
  - Consultorio Verónica Salem, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Consultorio Silvia Goso, Buenos Aires
  - Consultorio Mariana Butty, Buenos Aires
  - Consultorio Esteban Azumendi, Buenos Aires
- Costa Rica (2):
  - Consultorio Ileana Morera Vargas, Alajuela
  - Consultorio Creciendo en Pareja, San José
- Clínica Humanamente Guatemala, Guatemala City, Guatemala
- Mexico (5):
  - Consulta Mónica Díaz Cayeros, Cancún, Quintana Roo
  - Consulta Alfonso Villareal, Mérida, Yucatán
  - Consulta Ali Barbosa, Mérida, Yucatán
  - Consulta Gerardo Vázquez, Mexico City
  - Consulta Cecilia Paredes, Mexico City
- Spain (4):
  - Consulta Itziar Arana, El Escorial, Madrid
  - Centro de Orientación y Mediación Familiar Coordenadas, Málaga
  - Gabinete de Terapia de Pareja de Zaragoza, Zaragoza
  - Centro Vitae Psicología, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez-Gonzalez M, Anderson S, Osorio A, Lafontaine MF, Greenman PS, Calatrava M, Andrade D, Lybbert R, Martinez-Diaz P, Steffen P, de Irala J, Sandberg J. Efficacy of Emotionally Focused Therapy among Spanish-speaking couples: study protocol of a randomized clinical trial in Argentina, Costa Rica, Guatemala, Mexico, and Spain. Trials. 2022 Oct 22;23(1):891. doi: 10.1186/s13063-022-06831-7. PMID 36273180

DOCUMENTS (1):
  • Informed Consent Form (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04277325/ICF_001.pdf